CLINICAL TRIAL: NCT03150810
Title: A Phase 1b Study to Assess the Safety, Tolerability and Clinical Activity of BGB-290 in Combination With Temozolomide (TMZ) in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study to Assess Safety, Tolerability and Clinical Activity of BGB-290 in Combination With Temozolomide (TMZ) in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Collaborators: Myriad Genetics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-290-103; 2017-001553-14 (EudraCT Number)
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
Keywords: Ovarian cancer; Triple negative breast cancer; Small cell lung cancer; Gastric cancer; temozolomide; BGB-290; antineoplastic agents; alkylating, alkylating agents,; Poly (ADP-ribose) polymerase inhibitors; enzyme inhibitors; Head and neck cancer; Esophageal cancer; Soft tissue sarcoma; Non small cell lung cancer; pamiparib
MeSH Terms: conditions — Ovarian Neoplasms; Triple Negative Breast Neoplasms; Small Cell Lung Carcinoma; Stomach Neoplasms; Head and Neck Neoplasms; Esophageal Neoplasms; Sarcoma; Carcinoma, Non-Small-Cell Lung | interventions — pamiparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 milligrams (mg) (Days 1-7) (Experimental): Pamiparib 60 mg twice daily on Days 1 to 28 in combination with pulse dosing of TMZ 40 mg once daily on Days 1 to 7 within a 28-day cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) (Experimental): Pamiparib 60 mg twice daily on Days 1 to 28 in combination with pulse dosing of TMZ 60 mg once daily on Days 1 to 7 within a 28-day cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) (Experimental): Pamiparib 60 mg twice daily on Days 1 to 28 in combination with pulse dosing of TMZ 80 mg once daily on Days 1 to 7 within a 28-day cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) (Experimental): Pamiparib 60 mg twice daily on Days 1 to 28 in combination with pulse dosing of TMZ 100 mg once daily on Days 1 to 7 within a 28-day cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) (Experimental): Pamiparib 60 mg twice daily on Days 1 to 28 in combination with pulse dosing of TMZ 120 mg once daily on Days 1 to 7 within a 28-day cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) (Experimental): Pamiparib 60 mg twice daily on Days 1 to 28 in combination with pulse dosing of TMZ 40 mg once daily on Days 1 to 14 within a 28-day cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) (Experimental): Pamiparib 60 mg twice daily in combination with TMZ 20 mg once daily administered continuously on Days 1 to 28 within a 28-day cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28) (Experimental): Pamiparib 60 mg twice daily in combination with TMZ 40 mg once daily administered continuously on Days 1 to 28 within a 28-day cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- Dose Expansion: Gastric Cancer (Experimental): Participants with gastric or gastroesophageal junction cancer received TMZ 60 mg administered on Days 1 to 7 in combination with pamiparib 60 mg twice daily on Days 1 to 28 of each cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- Dose Expansion: Ovarian Cancer (Experimental): Participants with ovarian cancer, fallopian cancer, or primary peritoneal cancer received TMZ 60 mg administered on Days 1 to 7 in combination with pamiparib 60 mg twice daily on Days 1 to 28 of each cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- Dose Expansion: SCLC (Experimental): Participants with Small Cell Lung Cancer (SCLC) received TMZ 60 mg administered on Days 1 to 7 in combination with pamiparib 60 mg twice daily on Days 1 to 28 of each cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- Dose Expansion: TNBC (Experimental): Participants with triple negative breast cancer (TNBC) received TMZ 60 mg administered on Days 1 to 7 in combination with pamiparib 60 mg twice daily on Days 1 to 28 of each cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- Dose Expansion: Other HRD+ Cancers (Experimental): Participants with non-small cell lung cancer (NSCLC), esophageal cancer, squamous head and neck cancer, or soft tissue sarcomas whose tumors are homologous recombination deficiency (HRD)+ received TMZ 60 mg administered on Days 1 to 7 in combination with pamiparib 60 mg twice daily on Days 1 to 28 of each cycle
  Interventions: Drug: Pamiparib; Drug: Temozolomide

INTERVENTIONS:
Drug: Pamiparib — Administered by mouth as a capsule twice daily
  Other Names: BGB-290
Drug: Temozolomide — TMZ at various doses administered by mouth as a capsule once daily.
  Other Names: TMZ; temodar

SUMMARY:
The primary objective of this study was to determine the safety and tolerability of pamiparib, the maximum tolerated dose (MTD) or maximum administered dose (MAD) for pamiparib combined with TMZ, to select the recommended Phase 2 dose (RP2D) and schedule of pamiparib in combination with TMZ, and to determine the antitumor activity of pamiparib in combination with TMZ.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥18 years old with advanced or metastatic stage solid tumors
2. Eastern Cooperative Oncology Group (ECOG) status ≤ 1
3. Have disease either evaluable (dose-escalation cohort) or measurable (dose-escalation and -expansion cohorts) per RECIST V1.1, except for prostate cancer participants
4. Agree to provide archival tumor tissue
5. Additional inclusion criteria for dose expansion cohorts:

   * Participants with homologous recombination deficiency (HRD+) or known BRCA mutant ovarian cancer Previously received at least one line of platinum-containing therapy in the advanced or metastatic setting and No progression or recurrent disease within 6 months from last platinum-containing regimen.
   * Participants with HRD+ or known BRCA mutant triple-negative breast cancer Up to one prior platinum-containing treatment in any treatment setting and up to 3 prior lines of therapy in the advanced or metastatic setting
   * Participants with HRD+ or known BRCA mutant prostate cancer Chemotherapy-naïve or previously received up to two taxane-based chemotherapy regimens, with documented prostate cancer progression
   * Participants with small cell lung cancer and gastric cancer, previously received ≤ 2 prior lines of therapy
   * Other HRD+ solid tumors of multiple indications

Key Exclusion Criteria: All participants

1. Prior treatment with a poly adenosine diphosphate-ribose polymerase (PARP) inhibitor.
2. Refractory to platinum-based therapy (dose-expansion cohort).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (22):
- United States (7):
  - Start Midwest, Grand Rapids, Michigan
  - Washington University in St Louis, St Louis, Missouri
  - Mount Sinai Prime, New York, New York
  - Montefiore Medical Park At Eastchester Einstein Campus, The Bronx, New York
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Texas Oncology (Loop) Usor, Dallas, Texas
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Chris Obrien Lifehouse, Camperdown, New South Wales
  - Saint Vincents Hospital Sydney, Darlinghurst, New South Wales
  - Icon Cancer Centre South Brisbane, South Brisbane, Queensland
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
- Spain (7):
  - Hospital Universitario Vall Dhebron, Barcelona
  - Ico H Duran I Reynals, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Start Madrid Fundacion Jimenez Diaz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Virgen de La Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Northern Centre For Cancer Care, High Heaton
  - University College Hospital, London
  - Sarah Cannon Research Institute Uk, London

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in multiple study centers in Australia, Europe, and North America.
Groups:
- Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7): Pamiparib 60 mg twice daily on Days 1 to 28 in combination with pulse dosing of TMZ 40 mg once daily on Days 1 to 7 within a 28-day cycle
Period: Overall Study
Arm/Group | Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) | Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28) | Dose Expansion: Gastric Cancer | Dose Expansion: Ovarian Cancer | Dose Expansion: SCLC | Dose Expansion: TNBC | Dose Expansion: Other HRD+ Cancers
Started | 4 | 13 | 9 | 3 | 3 | 14 | 14 | 6 | 21 | 4 | 22 | 1 | 25
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 13 | 9 | 3 | 3 | 14 | 14 | 6 | 21 | 4 | 22 | 1 | 25
Not completed — Death | 4 | 8 | 7 | 2 | 2 | 10 | 8 | 6 | 18 | 3 | 19 | 1 | 19
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 1
Not completed — Sponsor Decision | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site withdrawal from study | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Hospice | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant relocated abroad. | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Transferred care to oncologist | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Expansion: Gastric Cancer: Participants with gastric or gastroesophageal junction cancer received TMZ 60 mg once daily administered on Days 1 to 7 in combination with pamiparib 60 mg twice daily on Days 1 to 28 of each cycle
- Dose Expansion: Ovarian Cancer: Participants with ovarian cancer, fallopian cancer, or primary peritoneal cancer received TMZ 60 mg once daily administered on Days 1 to 7 in combination with pamiparib 60 mg twice daily on Days 1 to 28 of each cycle
- Dose Expansion: SCLC: Participants with Small Cell Lung Cancer (SCLC) received TMZ 60 mg once daily administered on Days 1 to 7 in combination with pamiparib 60 mg twice daily on Days 1 to 28 of each cycle
- Dose Expansion: TNBC: Participants with triple negative breast cancer (TNBC) received TMZ 60 mg once daily administered on Days 1 to 7 in combination with pamiparib 60 mg twice daily on Days 1 to 28 of each cycle
- Dose Expansion: Other HRD+ Cancers: Participants with non-small cell lung cancer (NSCLC), esophageal cancer, squamous head and neck cancer, or soft tissue sarcomas whose tumors are homologous recombination deficiency (HRD)+ received TMZ 60 mg once daily administered on Days 1 to 7 in combination with pamiparib 60 mg twice daily on Days 1 to 28 of each cycle
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) | Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28) | Dose Expansion: Gastric Cancer | Dose Expansion: Ovarian Cancer | Dose Expansion: SCLC | Dose Expansion: TNBC | Dose Expansion: Other HRD+ Cancers | Total
Number analyzed (Participants) | 4 | 13 | 9 | 3 | 3 | 14 | 14 | 6 | 21 | 4 | 22 | 1 | 25 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (6.19) | 58.0 (10.52) | 72.3 (6.22) | 60.3 (10.69) | 65.7 (13.80) | 66.7 (10.21) | 66.9 (9.96) | 66.7 (8.31) | 58.8 (14.68) | 59.3 (2.22) | 61.9 (8.33) | 31.0 (NA) — Not Estimable | 58.1 (8.28) | 62.0 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 5 | 2 | 1 | 6 | 7 | 2 | 8 | 4 | 8 | 1 | 10 | 64
  Male | 1 | 6 | 4 | 1 | 2 | 8 | 7 | 4 | 13 | 0 | 14 | 0 | 15 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 0 | 0 | 1 | 5 | 1 | 1 | 1 | 0 | 0 | 0 | 12
  Not Hispanic or Latino | 4 | 11 | 7 | 2 | 3 | 11 | 8 | 4 | 18 | 3 | 18 | 1 | 20 | 110
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 0 | 4 | 0 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 10
  White | 4 | 10 | 9 | 2 | 1 | 7 | 8 | 5 | 18 | 2 | 18 | 1 | 20 | 105
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 3 | 5 | 0 | 1 | 1 | 4 | 0 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT is defined as one of the following toxicities occurring during the DLT assessment window:
  Grade ≥3 non-hematologic, non-hepatic major organ adverse event (AE) Grade 4 neutropenia lasting >7 days Grade ≥3 febrile neutropenia Grade 3 thrombocytopenia with clinically significant bleeding Grade 4 thrombocytopenia lasting > 3 days and requiring transfusion, or any decreased platelet count <15,000/mm3/ <15.0 x 109/L Grade ≥4 anemia Grade ≥3 total bilirubin or hepatic transaminases (ALT or AST)
Time Frame: From first dose of study drug(s) to 28 days post-dose (up to approximately 1 year and 6 months)
Population: The dose-escalation safety analysis set comprised all dose-escalation phase participants who received pamiparib and/or TMZ.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) | Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28)
Number analyzed (Participants) | 4 | 13 | 9 | 3 | 3 | 14 | 14 | 6
Participants | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including laboratory values, vital signs, physical examination findings, and electrocardiogram results, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v4.03
Time Frame: From the first dose of study drug(s) to 30 days after the last dose; up to approximately 5 years and 10 months
Population: The Safety Analysis Set included all participants who received any dose of pamiparib and/or TMZ.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) | Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28) | Dose Expansion: Gastric Cancer | Dose Expansion: Ovarian Cancer | Dose Expansion: SCLC | Dose Expansion: TNBC | Dose Expansion: Other HRD+ Cancers
Number analyzed (Participants) | 4 | 13 | 9 | 3 | 3 | 14 | 14 | 6 | 21 | 4 | 22 | 1 | 25
Participants
  Participants With At Least 1 TEAE | 4 | 13 | 9 | 3 | 3 | 14 | 14 | 6 | 20 | 4 | 22 | 1 | 24
  Participants with Serious TEAEs | 1 | 4 | 1 | 2 | 2 | 5 | 5 | 0 | 9 | 3 | 9 | 0 | 9

3. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants who have a best overall response (BOR) of complete response (CR) or partial response (PR) based on investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, where BOR is defined as the best response recorded from the first postbaseline tumor assessment until data cutoff date, disease progression or start of new anticancer treatment.
Time Frame: Up to approximately 5 years and 10 months
Population: The Efficacy Analysis Set included all participants who were in the safety analysis set, had measurable disease at baseline and had at least one postbaseline tumor assessment unless discontinued treatment due to clinical progression or death prior to tumor assessment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) | Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28) | Dose Expansion: Gastric Cancer | Dose Expansion: Ovarian Cancer | Dose Expansion: SCLC | Dose Expansion: TNBC | Dose Expansion: Other HRD+ Cancers
Number analyzed (Participants) | 3 | 12 | 8 | 2 | 2 | 14 | 13 | 4 | 19 | 4 | 20 | 1 | 25
percentage of participants | 0.0 [0.0 to 63.2] | 16.7 [3.0 to 43.8] | 25.0 [4.6 to 60.0] | 0.0 [0.0 to 77.6] | 0.0 [0.0 to 77.6] | 21.4 [6.1 to 46.6] | 0.0 [0.0 to 20.6] | 25.0 [1.3 to 75.1] | 0.0 [0.0 to 14.6] | 50.0 [9.8 to 90.2] | 15.0 [4.2 to 34.4] | 100.0 [5.0 to 100.0] | 8.0 [1.4 to 23.1]

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Pamiparib
Description: Pamiparib pharmakokinetic (PK) parameters were assessed in the first 20 participants enrolled in the dose escalation phase after a single dose on Day -2 and at steady state in combination with TMZ on Day 15.
Time Frame: 2 days before Cycle 1 Day 1 (Day -2) at predose, 30 min, 1, 2, 4, 6, 24, and 48 hours after dosing, and on Cycle 1 Day 15 at predose, 1, 2, and 4 hours postdose (each cycle is 28 days)
Population: The pamiparib pharmacokinetic analysis included the first 20 participants enrolled in the dose escalation phase; per the prespecified analysis, participants were analyzed in one group, regardless of dose of TMZ they received. Only 13 participants had data available for calculation of Cmax on Day 15.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Pamiparib: The first 20 participants enrolled in the dose-escalation phase received a single dose of 60 mg pamiparib on Day -2, prior to initiating twice daily dosing with 60 mg pamiparib and TMZ per assigned treatment group on Day 1.
Arm/Group | Pamiparib
Number analyzed (Participants) | 20
ng/mL
  Day -2 | 1945.31 (25)
  Cycle 1 Day 15: number analyzed (Participants) | 13
  Cycle 1 Day 15 | 3796.06 (33)

5. Secondary Outcome: Plasma Trough Concentrations of Pamiparib (Ctrough)
Time Frame: Cycle 1 Day 15 predose
Population: The pamiparib pharmacokinetic analysis included the first 20 participants enrolled in the dose escalation phase; per the prespecified analysis, participants were analyzed in one group, regardless of dose of TMZ they received. Only 14 participants had data available for calculation of Ctrough on Day 15.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pamiparib
Number analyzed (Participants) | 14
ng/mL | 2335.6 (76)

6. Secondary Outcome: Time to Reach Cmax (Tmax) of Pamiparib
Time Frame: 2 days before Cycle 1 Day 1 (Day -2) at predose, 30 min, 1, 2, 4, 6, 24, and 48 hours after dosing, and on Cycle 1 Day 15 at predose, 1, 2, and 4 hours postdose.
Population: The pamiparib pharmacokinetic analysis included the first 20 participants enrolled in the dose escalation phase; per the prespecified analysis, participants were analyzed in one group, regardless of dose of TMZ they received. Only 13 participants had data available for calculation of Tmax on Day 15.
Measure: Median (Full Range); unit: hours
Arm/Group | Pamiparib
Number analyzed (Participants) | 20
hours
  Day -2 | 2.00 [1.00 to 23.92]
  Cycle 1 Day 15: number analyzed (Participants) | 13
  Cycle 1 Day 15 | 1.83 [0.83 to 2.17]

7. Secondary Outcome: Area Under the Curve From Time 0 to 4 Hours (AUC0-4h) of Pamiparib
Time Frame: 2 days before Cycle 1 Day 1 (Day -2) at predose, 30 min, 1, 2, and 4 hours after dosing, and on Cycle 1 Day 15 at predose, 1, 2, and 4 hours postdose.
Population: The pamiparib pharmacokinetic analysis included the first 20 participants enrolled in the dose escalation phase; per the prespecified analysis participants were analyzed in one group, regardless of dose of TMZ they received. Only 8 participants had available data to calculate AUC0-4 on Day 15.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pamiparib
Number analyzed (Participants) | 20
h*ng/mL
  Day -2 | 4646.4 (45)
  Cycle 1 Day 15: number analyzed (Participants) | 8
  Cycle 1 Day 15 | 11119.5 (41)

8. Secondary Outcome: Area Under the Curve From Time 0 to Infinity (AUC0-inf) of Pamiparib
Time Frame: 2 days before Cycle 1 Day 1 (Day -2) at predose, 30 min, 1, 2, 4, 6, 24, and 48 hours after dosing
Population: The pamiparib pharmacokinetic analysis included the first 20 participants enrolled in the dose escalation phase; AUC0-inf could only be calculated for 15 participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pamiparib
Number analyzed (Participants) | 15
h*ng/mL | 25287.0 (50)

9. Secondary Outcome: Terminal Elimination Half-life (t1/2) of Pamiparib
Time Frame: 2 days before Cycle 1 Day 1 (Day -2) at predose, 30 min, 1, 2, 4, 6, 24, and 48 hours after dosing (each cycle is 28 days)
Population: The pamiparib pharmacokinetic analysis included the first 20 participants enrolled in the dose escalation phase; Only 17 participants had data available to calculate T1/2.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Pamiparib
Number analyzed (Participants) | 17
hours | 11.82 [5.94 to 33.58]

10. Secondary Outcome: Apparent Clearance (CL/F) of Pamiparib
Time Frame: as for outcome 9
Population: The pamiparib pharmacokinetic analysis included the first 20 participants enrolled in the dose escalation phase; Only 15 participants had data available to calculate CL/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Pamiparib
Number analyzed (Participants) | 15
L/h | 2.37 (50)

11. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/F) of Pamiparib
Time Frame: as for outcome 9
Population: The pamiparib pharmacokinetic analysis included the first 20 participants enrolled in the dose escalation phase; Only 15 participants had data available to calculate Vz/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Pamiparib
Number analyzed (Participants) | 15
liters | 38.14 (15)

12. Secondary Outcome: Plasma Concentration of Temozolomide (TMZ)
Time Frame: Predose (within 30 min prior to dose) and 1 hour post dose on Cycle 1 Day 1 and Cycle 1 Day 7
Population: PK Analysis Set: includes participants who received any dose of TMZ and contributed at least one plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- TMZ 20 mg: Participants who received 20 mg TMZ orally once a day.
- TMZ 40 mg: Participants who received 40 mg TMZ orally once a day.
- TMZ 60 mg: Participants who received 60 mg TMZ orally once a day.
- TMZ 80 mg: Participants who received 80 mg TMZ orally once a day.
- TMZ 100 mg: Participants who received 100 mg TMZ orally once a day.
- TMZ 120 mg: Participants who received 120 mg TMZ orally once a day.
Arm/Group | TMZ 20 mg | TMZ 40 mg | TMZ 60 mg | TMZ 80 mg | TMZ 100 mg | TMZ 120 mg
Number analyzed (Participants) | 14 | 24 | 85 | 9 | 3 | 3
ng/mL
  C1D1 Predose: number analyzed (Participants) | 5 | 15 | 19 | 5 | 2 | 3
  C1D1 Predose | NA (NA) — All pre-dose concentrations noted as NA were below limit of quantitation | NA (NA) — All pre-dose concentrations noted as NA were below limit of quantitation | NA (NA) — All pre-dose concentrations noted as NA were below limit of quantitation | NA (NA) — All pre-dose concentrations noted as NA were below limit of quantitation | NA (NA) — All pre-dose concentrations noted as NA were below limit of quantitation | NA (NA) — All pre-dose concentrations noted as NA were below limit of quantitation
  C1D1 Postdose 1H: number analyzed (Participants) | 7 | 15 | 17 | 5 | 2 | 3
  C1D1 Postdose 1H | 322.8 (35) | 601.3 (68) | 822.3 (74) | 1366.1 (46) | 1157.9 (123) | 1464.5 (31)
  C1D7 Predose: number analyzed (Participants) | 5 | 13 | 13 | 3 | 0 | 3
  C1D7 Predose | NA (NA) — All pre-dose concentrations noted as NA were below limit of quantitation | NA (NA) — All pre-dose concentrations noted as NA were below limit of quantitation | NA (NA) — All pre-dose concentrations noted as NA were below limit of quantitation | NA (NA) — All pre-dose concentrations noted as NA were below limit of quantitation |  | NA (NA) — All pre-dose concentrations noted as NA were below limit of quantitation
  C1D7 Postdose 1H: number analyzed (Participants) | 5 | 13 | 12 | 3 | 1 | 3
  C1D7 Postdose 1H | 340.9 (86) | 636.7 (57) | 761.1 (103) | 1959.8 (40) | 1520.0 | 1775.6 (71)

13. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with BOR of CR, PR, or stable disease (SD) based on investigator assessment using RECIST v1.1.
Time Frame: Up to approximately 5 years and 10 months
Population: Efficacy Analysis Set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) | Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28) | Dose Expansion: Gastric Cancer | Dose Expansion: Ovarian Cancer | Dose Expansion: SCLC | Dose Expansion: TNBC | Dose Expansion: Other HRD+ Cancers
Number analyzed (Participants) | 3 | 12 | 8 | 2 | 2 | 14 | 13 | 4 | 19 | 4 | 20 | 1 | 25
percentage of participants | 33.3 [1.7 to 86.5] | 91.7 [66.1 to 99.6] | 75.0 [40.0 to 95.4] | 100.0 [22.4 to 100] | 50.0 [2.5 to 97.5] | 42.9 [20.6 to 67.5] | 53.8 [28.7 to 77.6] | 75.0 [24.9 to 98.7] | 42.1 [23.0 to 63.2] | 75.0 [24.9 to 98.7] | 75.0 [54.4 to 89.6] | 100.0 [5.0 to 100] | 52.0 [34.1 to 69.5]

14. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the date of the earliest documented CR or PR (that is subsequently confirmed) to disease progression or death due to any cause, whichever occurs earlier, based on investigator assessment using RECIST v1.1. Only responders will be included in the assessment.
Time Frame: Up to approximately 5 years and 10 months
Population: Efficacy Analysis Set
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) | Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28) | Dose Expansion: Gastric Cancer | Dose Expansion: Ovarian Cancer | Dose Expansion: SCLC | Dose Expansion: TNBC | Dose Expansion: Other HRD+ Cancers
Number analyzed (Participants) | 0 | 2 | 2 | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 3 | 1 | 2
months |  | 13.0 [NA to NA] — NA = Not estimable due to insufficient number of participants with events | 6.4 [5.5 to NA] — NA = Not estimable due to insufficient number of participants with events |  |  | 9.2 [7.7 to NA] — NA = Not estimable due to insufficient number of participants with events |  | 3.7 [NA to NA] — NA = Not estimable due to insufficient number of participants with events |  | 5.4 [4.9 to NA] — NA = Not estimable due to insufficient number of participants with events | 3.8 [3.2 to NA] — NA = Not estimable due to insufficient number of participants with events | 11.0 [NA to NA] — NA = Not estimable due to insufficient number of participants with events | NA [7.4 to NA] — NA = Not estimable due to insufficient number of participants with events

15. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time (months) from the date of the first dose of combination treatment to disease progression or death due to any cause, whichever occurs first, based on investigator assessment using RECIST v1.1
Time Frame: Up to approximately 5 years and 10 months)
Population: Efficacy Analysis Set
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) | Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28) | Dose Expansion: Gastric Cancer | Dose Expansion: Ovarian Cancer | Dose Expansion: SCLC | Dose Expansion: TNBC | Dose Expansion: Other HRD+ Cancers
Number analyzed (Participants) | 3 | 12 | 8 | 2 | 2 | 14 | 13 | 4 | 19 | 4 | 20 | 1 | 25
months | 2.0 [1.2 to NA] — NA = Not estimable due to insufficient number of participants with events | 5.6 [2.7 to 22] | 5.3 [1.8 to 7.5] | NA [4.5 to NA] — NA = Not estimable due to insufficient number of participants with events | NA [1.8 to NA] — NA = Not estimable due to insufficient number of participants with events | 2.8 [1.7 to 3.7] | 3.1 [1.7 to 3.9] | 3.5 [1.1 to NA] — NA = Not estimable due to insufficient number of participants with events | 1.9 [1.7 to 3.3] | 6.4 [2.6 to NA] — NA = Not estimable due to insufficient number of participants with events | 3.5 [2.3 to 4.1] | 14.8 [NA to NA] — NA = Not estimable due to insufficient number of participants with events | 2.6 [1.9 to 3.6]

16. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of the first dose of combination treatment to death due to any cause.
Time Frame: Up to approximately 5 years and 10 months
Population: The Safety Analysis Set included all participants who received any dose of pamiparib and/or TMZ.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) | Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28) | Dose Expansion: Gastric Cancer | Dose Expansion: Ovarian Cancer | Dose Expansion: SCLC | Dose Expansion: TNBC | Dose Expansion: Other HRD+ Cancers
Number analyzed (Participants) | 4 | 13 | 9 | 3 | 3 | 14 | 14 | 6 | 21 | 4 | 22 | 1 | 25
months | 7.6 [2.2 to NA] — NA = Not estimable due to insufficient number of events | 14.8 [8.4 to NA] — NA = Not estimable due to insufficient number of events | 12.7 [9.4 to NA] — NA = Not estimable due to insufficient number of events | 12.4 [4.5 to NA] — NA = Not estimable due to insufficient number of events | 12.3 [4.2 to NA] — NA = Not estimable due to insufficient number of events | 6.3 [3.4 to 31.8] | 13.9 [8.0 to NA] — NA = Not estimable due to insufficient number of events | 8.2 [1.1 to 12.7] | 6.6 [3.8 to 9.9] | 21.2 [11.1 to NA] — NA = Not estimable due to insufficient number of events | 7.7 [4.1 to 13.1] | 19.4 [NA to NA] — NA = Not estimable due to insufficient number of events | 9.8 [7.6 to 11.7]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events (AEs): From the first dose of study drug(s) to 30 days after the last dose; up to approximately 5 years and 10 months
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events include all randomized participants who received ≥ 1 dose of any study treatment
  AEs are defined as events that had an onset date or a worsening in severity from baseline (pretreatment) on or after the first dose of study treatment up to 30 days following study treatment discontinuation or initiation of a new anticancer therapy, whichever occurred first.
Arm/Group | Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) | Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28) | Dose Expansion: Gastric Cancer | Dose Expansion: Ovarian Cancer | Dose Expansion: SCLC | Dose Expansion: TNBC | Dose Expansion: Other HRD+ Cancers
All-Cause Mortality (participants affected / at risk) | 4/4 | 8/13 | 7/9 | 2/3 | 2/3 | 10/14 | 8/14 | 6/6 | 18/21 | 3/4 | 19/22 | 1/1 | 19/25
Serious Adverse Events (participants affected / at risk) | 1/4 | 4/13 | 1/9 | 2/3 | 2/3 | 5/14 | 5/14 | 0/6 | 9/21 | 3/4 | 9/22 | 0/1 | 9/25
Other Adverse Events (participants affected / at risk) | 4/4 | 13/13 | 9/9 | 3/3 | 3/3 | 14/14 | 14/14 | 6/6 | 20/21 | 4/4 | 22/22 | 1/1 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7) (N=4) | Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) (N=13) | Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) (N=9) | Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) (N=3) | Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) (N=3) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) (N=14) | Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) (N=14) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28) (N=6) | Dose Expansion: Gastric Cancer (N=21) | Dose Expansion: Ovarian Cancer (N=4) | Dose Expansion: SCLC (N=22) | Dose Expansion: TNBC (N=1) | Dose Expansion: Other HRD+ Cancers (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Right-to-left cardiac shunt (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Precerebral artery embolism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Pamiparib + Temozolomide (TMZ) 40 mg (Days 1-7) (N=4) | Dose Escalation: Pamiparib + TMZ 60 mg (Days 1-7) (N=13) | Dose Escalation: Pamiparib + TMZ 80 mg (Days 1-7) (N=9) | Dose Escalation: Pamiparib + TMZ 100 mg (Days 1-7) (N=3) | Dose Escalation: Pamiparib + TMZ 120 mg (Days 1-7) (N=3) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-14) (N=14) | Dose Escalation: Pamiparib + TMZ 20 mg (Days 1-28) (N=14) | Dose Escalation: Pamiparib + TMZ 40 mg (Days 1-28) (N=6) | Dose Expansion: Gastric Cancer (N=21) | Dose Expansion: Ovarian Cancer (N=4) | Dose Expansion: SCLC (N=22) | Dose Expansion: TNBC (N=1) | Dose Expansion: Other HRD+ Cancers (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 8 (11) | 5 (8) | 2 (8) | 3 (4) | 10 (15) | 6 (10) | 3 (4) | 12 (15) | 2 (4) | 13 (18) | 1 (4) | 16 (25)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (8) | 3 (5) | 2 (8) | 3 (4) | 5 (16) | 3 (4) | 1 (1) | 5 (6) | 3 (3) | 6 (7) | 1 (5) | 5 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 5 (10) | 4 (5) | 1 (6) | 3 (9) | 7 (15) | 1 (1) | 2 (2) | 6 (6) | 2 (5) | 6 (12) | 0 (0) | 3 (4)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 1 (1) | 5 (6) | 2 (2) | 6 (6) | 0 (0) | 4 (8)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (5) | 3 (4) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 2 (2) | 5 (9) | 2 (4) | 3 (6) | 1 (1) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 9 (12) | 5 (5) | 2 (2) | 2 (2) | 5 (6) | 6 (8) | 4 (4) | 12 (14) | 4 (4) | 12 (20) | 1 (1) | 7 (10)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Saliva altered (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Tongue pigmentation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 4 (10) | 2 (2) | 1 (1) | 10 (15) | 2 (2) | 7 (12) | 0 (0) | 4 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 5 (7)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 9 (10) | 5 (5) | 1 (2) | 1 (1) | 10 (10) | 4 (6) | 2 (2) | 12 (13) | 3 (3) | 13 (19) | 0 (0) | 7 (9)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Sluggishness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device occlusion (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 2 (2) | 4 (5) | 0 (0) | 7 (11) | 0 (0) | 8 (15)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 2 (2) | 3 (7) | 2 (2) | 5 (5) | 1 (1) | 9 (14) | 1 (6) | 8 (8)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 5 (8) | 1 (1) | 8 (8) | 3 (3) | 11 (12) | 0 (0) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 4 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Areflexia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 4 (6) | 1 (1) | 2 (2)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 0 (0) | 4 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (4) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Xanthoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Capillary fragility (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights

DOCUMENTS (2):
  • Study Protocol (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT03150810/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT03150810/SAP_001.pdf